CLINICAL TRIAL: NCT05118945
Title: Observational Study on the Use of the Insulin Pump Tandem X:2 With Control IQ Algorithm - Update
Brief Title: Study on the Use of the Insulin Pump Tandem X:2 With Control IQ Algorithm - Update
Acronym: UNIQUE
Status: Completed | Type: Observational
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Responsible Party: Sponsor
Other Study IDs: Unique_1_2021
Record Dates: First submitted 2021-10-12; First posted 2021-11-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes; Insulin Therapy
Keywords: paediatrics; type 1 diabetes; closed loop; CSII (Continuous Subcutaneous Insulin Infusion)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SWITCH group: Change from Basal IQ to Control IQ: The patients of the SWITCH group used the X:s insulin pump with the "Basal IQ" algorithm until the start of the study and switched to the "Control IQ" algorithm at study start.
  Interventions: Device: Insulin pump Tandem: t:slim X2
- START group: Change from conservative therapy to Control IQ: The patients of the START group have a conservative Insulin therapy (MDI = multiple daily injections or CSII = Continuous subcutaneous insulin infusion) until the start of the study, but will switched to the "Control IQ" algorithm at study start.
  Interventions: Device: Insulin pump Tandem: t:slim X2

INTERVENTIONS:
Device: Insulin pump Tandem: t:slim X2 — Insulin pump with Hybrid-Closed Loop - Modus. The insulin pump t:slim X2 from the manufacturer Tandem, in cooperation with the glucose sensor DexCom G6, has the option of using an algorithm called "control IQ", which controls the insulin delivery semi-automatically by means of an MPC algorithm. For this purpose, the insulin basal delivery can be increased or decreased by the system. Furthermore, automatic bolus deliveries, which are possible in the amount of up to 60% of a manual correction, can be delivered.
  Other Names: Insulin pump Tandem: t:slim X2 with Control IQ

SUMMARY:
The aim of this observational clinical trial is to obtain data on the safety, efficacy and satisfaction of the Tandem T:Slim X:2 Pump System in patients with type 1 diabetes.

DETAILED DESCRIPTION:
This is a non-randomized, non-blinded, prospective, observational single-center study, enrolling 2x 25 subjects in two cohorts (25 subjects in SWITCH group and 25 subjects in START group) with diabetes mellitus for up to 12 weeks. The study will evaluate the effectiveness of the insulin therapy with the pump system Tandem t:slim X:2 with the special algorithm "Control IQ" in comparison to each other. The test system including the Control IQ software will provide an Hybrid-Closed loop - Modus, which can predict the future tissue glucose value and continuously adjust the insulin infusion according to need. The aim is to keep the glucose value permanently within the target range and to avoid hypoglycaemia or hyperglycaemia.

Group START starts from any other diabetes therapy (MDI, PLGM (=Predictive Low Glucose Suspend), SaP (=Sensor augmented Pump)) directly to T:Slim pump with control IQ; group SWITCH switches from former use of T:slim with Basal IQ.

The study includes two visits only (start and end). At the beginning all patients have to complete questionnaires, and the data of the glucose sensor are read out and the metric data are determined and laid down.

Depending on the previous form of therapy, the patients are assigned to the corresponding cohort. All participants and parents, regardless of which cohort, receive a technical briefing from the study team as well as training on how to use the new system or algorithm. Subsequently, the system will be applied in everyday life in the coming weeks. After 12 weeks (end of study), the insulin pump is read out and the questionnaire on satisfaction with the device is filled out again.

After the end of the study, the patients participate in standard medical care as before.

ELIGIBILITY:
Inclusion Criteria:

1. signed informed consent
2. type 1 diabetes
3. Age >6 years
4. at least 10 IE daily total Insulin dose and 25 kg Body weight
5. Group SWITCH: already user of t:slim X2 with Basal IQ
6. Group START: Granting of the insulin pump t:slim X2 and DexCom G6 by the health insurance

Exclusion Criteria:

1.Refusal of participation by the participant or a parent

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients over 6 years of age with type 1 Diabetes and Insulin therapy (MDI or CSII).
  The START group is heterogeneous, but it should be ensured that all patients in the start group do not use a close loop system so far.
  Furthermore, a maximum of 30 % of the patients in the START group should use the same pump system to ensure that the weighting of a single pump system does not become too strong.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Time in glucose range 70 - 180mg/dl (%) | 12 weeks
  Both groups are evaluated together. Comparison of the time (%) in the glucose range 70 - 180mg/dl of the last two weeks of the study with the time in the target range two weeks before the start of the study.

SECONDARY OUTCOMES:
user satisfaction assessed by disabkids questionnaire for children and for parents | two weeks
  Comparison of both groups with regard to satisfaction via specific validated questionnaire at the start of the study
user satisfaction assessed by disabkids questionnaire for children and for parents | 12 weeks
  Evaluation of the satisfaction of users via specific validated questionnare at the beginning and the end of study
mean glucose level [mg/dl] | two weeks
  Comparison of the mean Glucose Level from glucose sensor [mg/dl] of the last two study weeks with the mean glucose Level two weeks before the start of the study.
mean glucose Level before study start [mg/dl] | two weeks
  Comparison of both groups concerning the mean glucose level of the two weeks before the start of the study.
mean daily insulin amount | 12 weeks
  Both groups are evaluated together. Comparison of the mean daily insulin amount (U/kgBW/d) (U/kgBW/d) of the last two study weeks with the insulin amount two weeks before the start of the study.
mean daily insulin amount before study start | two weeks
  Comparison of both groups concerning the mean daily insulin amount (U/kgBW/d) of the two weeks before the start of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Torben Biester, Dr., Principal Investigator — Hospital for Children and Adolescents AUF DER BULT
Locations (1):
- Hospital for Children and Adolescents AUF DER BULT, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No